CLINICAL TRIAL: NCT00353002
Title: A Comparison of Amethocaine Creams Versus Liposomal Lidocaine Cream as Pain Reliever Prior to Venipuncture in Children at the Paediatric Emergency Department.
Brief Title: A Comparison of Amethocaine Cream vs. Liposomal Lidocaine Cream for Venipuncture in Children.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R-06-266; LHRI IRF (Other Grant/Funding Number: LHRI)
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Pain
Keywords: Pain; Ametop; Liposomal Lidocaine; Venous cannulation
MeSH Terms: conditions — Pain | interventions — Tetracaine; Maxilene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Ametop (4% Amethocaine cream )
Drug: Maxilene (4% Liposomal Lidocaine)

SUMMARY:
All patients undergoing venepuncture or venous cannulation in pediatric emergency department will be treated with either Amethocaine, or Liposomal Lidocaine (4%) cream at the site of cannulation in order to determine the efficacy of these creams in controlling pain during procedures and to determine the success rate of these procedures.

DETAILED DESCRIPTION:
Children commonly require blood taking or placement of an intravenous line for both diagnosis and treatment during their visit to the emergency department. The distress from needle puncture is a particular issue in children. The development of needle phobia can subsequently adversely affect the well-being of the children and their relationship with the medical staff. Thus reduction of pain and distress would be beneficial to patients, parents, and medical personnel.

Amethocaine (tetracaine 4%) (Ametop) is another topical anaesthetic cream which was marketed in Canada over the last 10 years; it was developed by Dr. David Wollfson at Queen's University, Belfast, the cream is available in a 1.5g tube that delivers only 1 dose, at a cost of ($3.24). structurally it has an ester type bond (Para-amino benzoic acid) and is formulated as a free base to allow tetracaine to diffuse across the skin barrier and reach pain receptors (nociceptors) which are located below the stratum corneum (outer most layer of skin). It acts by inhibiting sodium ion flux across the axon membrane thus preventing the nociceptors from signalling pain to the central nervous system. The application time required for the cream is only 30 minutes, and it possesses an action time of 4 hours after removal from the skin. Also Amethocaine has a low risk for methemoglobinemia, therefore it can be used safely in neonatal period and the only disadvantage of Amethocaine cream is skin erythema due to vasodilatation effect.

Liposomal lidocaine 4% cream (Maxilene, RGR Pharma, Windsor, Ontario) is another anaesthetic cream that was launched recently in Canada in 2003. And 5 gm tube priced is 15 $. The liposome-encapsulated formulation protects the anesthetic from being metabolized too quickly (12) It has short onset of action and minimal vasoactive properties that minimize any potential interference with cannulation success, and it is not associated with methemoglobinemia.

As of yet, there has not been a study done in children in the Emergency Department setting comparing the efficacy and side effects of both Liposomal Lidocaine cream and Amethocaine cream. Thus, there is no evidence guiding the use of these agents in Paediatric Emergency care setting, Furthermore using these creams are not considered standard care for children in Canada, and the usual clinical practice in Canadian emergency departments is not to use local anesthesia creams before IV insertion or blood extraction.

Thus, if positive the results of this study could be directly applied to changing the care of children in acute and emergency care setting.

Both creams have shown considerable potential in alleviating procedure pain, but both creams can also cause skin effect, and thus may affect the success rate of these procedures. Therefore we would like to test the two creams to demonstrate the efficacy of these two creams in controlling pain. As Liposomal Lidocaine is believed to have fewer side and skin effects than Amethocaine, it's possible that the success rate may be better with Liposomal Lidocaine than with Amethocaine cream and thus would be preferred agent for use for children in the Emergency and acute care setting.

ELIGIBILITY:
Inclusion Criteria:

* All children age who are visiting the paediatric emergency department and need for IV cannulation or blood workup as part of their management. The need for IV placement or blood drawing will be based on the clinical evaluation of the child by experienced triage nursing personnel.

Exclusion Criteria:

* Lack of parental agreement
* Broken skin
* Known sensitivity to Amethocaine or Liposomal Lidocaine cream.
* Children with critical illness requiring immediate cannulation (e.g., sepsis, severe dehydration, Trauma)
* Children who are already receiving opioid analgesia or topical anesthesia.
* Children who have already participated in the study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2006-07 (Actual); Study Completion 2006-12

PRIMARY OUTCOMES:
Facial pain scale score of child during procedure | Immediate

SECONDARY OUTCOMES:
Compare local and systemic side effects of both creams | Within hour of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Rieder, MD PhD FRCPC, Principal Investigator — Children's Hospital of Western Ontario, University of Western Ontario; Khalid Alawi, MD FRCPC, Study Director — Children's Hospital of Western Ontario
Locations (1):
- Children's Hospital of Western Ontario, London, Ontario, Canada

REFERENCES:
- [Background] Browne J, Awad I, Plant R, McAdoo J, Shorten G. Topical amethocaine (Ametop) is superior to EMLA for intravenous cannulation. Eutectic mixture of local anesthetics. Can J Anaesth. 1999 Nov;46(11):1014-8. doi: 10.1007/BF03013194. PMID 10566919
- [Background] Choy L, Collier J, Watson AR. Comparison of lignocaine-prilocaine cream and amethocaine gel for local analgesia before venepuncture in children. Acta Paediatr. 1999 Sep;88(9):961-4. doi: 10.1080/08035259950168450. PMID 10519337
- [Background] Taddio A, Soin HK, Schuh S, Koren G, Scolnik D. Liposomal lidocaine to improve procedural success rates and reduce procedural pain among children: a randomized controlled trial. CMAJ. 2005 Jun 21;172(13):1691-5. doi: 10.1503/cmaj.045316. PMID 15967972
- [Background] Lawson RA, Smart NG, Gudgeon AC, Morton NS. Evaluation of an amethocaine gel preparation for percutaneous analgesia before venous cannulation in children. Br J Anaesth. 1995 Sep;75(3):282-5. doi: 10.1093/bja/75.3.282. PMID 7547043
- [Background] Bishai R, Taddio A, Bar-Oz B, Freedman MH, Koren G. Relative efficacy of amethocaine gel and lidocaine-prilocaine cream for Port-a-Cath puncture in children. Pediatrics. 1999 Sep;104(3):e31. doi: 10.1542/peds.104.3.e31. PMID 10469814
- [Background] Eichenfield LF, Funk A, Fallon-Friedlander S, Cunningham BB. A clinical study to evaluate the efficacy of ELA-Max (4% liposomal lidocaine) as compared with eutectic mixture of local anesthetics cream for pain reduction of venipuncture in children. Pediatrics. 2002 Jun;109(6):1093-9. doi: 10.1542/peds.109.6.1093. PMID 12042548
- [Background] Cereda CM, de Araujo DR, Brunetto GB, De Paula E. Liposomal prilocaine: preparation, characterization, and in vivo evaluation. J Pharm Pharm Sci. 2004 Jul 15;7(2):235-40. PMID 15367381
- [Background] Bucalo BD, Mirikitani EJ, Moy RL. Comparison of skin anesthetic effect of liposomal lidocaine, nonliposomal lidocaine, and EMLA using 30-minute application time. Dermatol Surg. 1998 May;24(5):537-41. doi: 10.1111/j.1524-4725.1998.tb04203.x. PMID 9598008
- [Background] Arrowsmith J, Campbell C. A comparison of local anaesthetics for venepuncture. Arch Dis Child. 2000 Apr;82(4):309-10. doi: 10.1136/adc.82.4.309. PMID 10735838
- [Background] Zempsky WT, Cravero JP; American Academy of Pediatrics Committee on Pediatric Emergency Medicine and Section on Anesthesiology and Pain Medicine. Relief of pain and anxiety in pediatric patients in emergency medical systems. Pediatrics. 2004 Nov;114(5):1348-56. doi: 10.1542/peds.2004-1752. PMID 15520120